CLINICAL TRIAL: NCT03103100
Title: Comparing Bupivacaine, Lidocaine, and a Combination of Bupivacaine and Lidocaine for Labor Epidural Activation: A Prospective, Randomized, Double-Blind Study
Brief Title: Comparing Bupivacaine, Lidocaine, and a Combination of Bupivacaine and Lidocaine for Labor Epidural Activation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mark Powell, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F140903008
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Labor Pain
Keywords: Local anesthetic; Labor epidural
MeSH Terms: conditions — Labor Pain | interventions — Lidocaine; Lidoderm; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 1% Lidocaine (Active Comparator): Patients randomized into the lidocaine group will receive 10 mL of 1% lidocaine
  Interventions: Drug: 1% Lidocaine
- 0.25% Bupivacaine (Active Comparator): Patients randomized into the bupivacaine group will receive 10 mL of 0.25% bupivacaine
  Interventions: Drug: 0.25% Bupivacaine
- Bupivacaine plus Lidocaine (Active Comparator): Patients randomized into the bupivacaine group will receive 5 mL of 0.25% bupivacaine and 5 mL of 1% lidocaine.
  Interventions: Drug: Bupivacaine plus Lidocaine

INTERVENTIONS:
Drug: 1% Lidocaine — 10 mL of 1% lidocaine
  Other Names: Lidoderm, Xylocaine, Recticare, Anecream,; Solarcaine, Anestacon, Cutiecaine, Lidocoll,
  Arms: 1% Lidocaine
Drug: 0.25% Bupivacaine — 10 mL of 0.25% bupivacaine
  Other Names: Marcaine and Sensorcaine
  Arms: 0.25% Bupivacaine
Drug: Bupivacaine plus Lidocaine — 5 mL of 1% lidocaine and 5 mL of 0.25% bupivacaine
  Other Names: Lidoderm, Xylocaine, Recticare, Anecream, Lmx4, Akten,; Marcaine and Sensorcaine
  Arms: Bupivacaine plus Lidocaine

SUMMARY:
This study will compare and determine the most ideal local anesthetic (LA) solution to activate a labor epidural: lidocaine, bupivacaine, or a combination of bupivacaine plus lidocaine.

DETAILED DESCRIPTION:
The most common and effective method for controlling labor pains is a local anesthetic (LA) infusion through a lumbar epidural. To achieve adequate pain control during the first stage of labor - onset of contractions to complete cervical dilation - nerve fibers up to the T10 dermatome must be anesthetized. When a patient is in active labor and an epidural catheter is placed, the anesthesiologist must activate the epidural by administering LA through the epidural to promote spread of the LA in the epidural space to anesthetize the nerve fibers involved in the conduction of labor pains. The ideal LA to achieve this goal is one that would allow for the fastest onset to achieve quick pain relief with the fewest side effects.

Two commonly used LA to provide labor analgesia are bupivacaine and lidocaine. When low concentrations - 0.25% bupivacaine and 1% lidocaine - are used for labor analgesia, both of these LA can be administered safely with very little concern of major adverse effects associated with LA toxicity. Given that there is limited and conflicting evidence for the usefulness of the bupivacaine and lidocaine mixture especially as it relates to labor epidural activation, we hope to readdress these questions in an effort to determine whether or not the LA combination offers any distinct advantage over the individual LA. The investigators intend to determine the time it takes to achieve an adequate level (T10) for labor analgesia, the total spread of local anesthetic, and the degree of motor block as these factors will be important in determining the most optimal LA solution to activate a labor epidural. With the results from this study, the investigators hope to recommend a LA solution that will allow for the fastest pain relief in the laboring mother with the fewest side effects.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients over the age of 19 who are scheduled for an induction of labor and request an epidural are eligible for the study

Exclusion Criteria:

* age <19
* allergy to the drug or drug class
* preexisting neuropathy
* history of back pain prior to pregnancy or history of back surgery
* history of chronic opioid use
* history of hypertension or hypertensive disorders of pregnancy
* congenital or acquired cardiac disease
* contraindication to epidural placement (patient refusal, severe coagulopathy, infection at site of epidural needle insertion, severe hypovolemia)

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy females admitted for induction of labor
Enrollment: 75 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F Powell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
Started | 25 | 25 | 25
Completed | 23 | 25 | 23
Not Completed | 2 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 25 | 75
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve an Adequate Epidural Level for Labor Analgesia
Description: time it takes to achieve a T10 dermatome level by pinprick. A T10 dermatome level is what is needed to control labor pain.
Time Frame: Baseline to 1 hour
Population: In the 1% lidocaine group, 1 participant experienced an adverse event and was removed from analysis and 1 participant was removed because they did not receive the study drug. In the bupivacaine plus lidocaine group 2 patients were removed because they did not receive the study drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
Number analyzed (Participants) | 23 | 25 | 23
minutes | 7.0 (3.9) | 11.0 (5.8) | 8.5 (4.6)

2. Secondary Outcome: Number of Patients Who Achieve Adequate Analgesia
Description: The number of patients who received an adequate epidural level of T10 or higher
Time Frame: Baseline to 1 hour
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
Number analyzed (Participants) | 23 | 25 | 23
Participants | 23 | 25 | 23

3. Secondary Outcome: Degree of Motor Block
Description: degree of motor block which means the amount of weakness in the legs experienced by the participants. this was determined by using the Bromage scale where 4 = greatest amount of motor block or muscle weakness and 0 = the least amount of motor block.
Time Frame: Baseline to 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Bromage Score
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
Number analyzed (Participants) | 23 | 25 | 23
Bromage Score | 2.0 (0.6) | 1.7 (1.0) | 1.9 (0.9)

4. Secondary Outcome: Number of Patients Who Experienced of Maternal Hypotension
Description: Number of patients who experienced maternal hypotension defined as a blood pressure (BP) >20% decline from baseline and need for vasopressor therapy
Time Frame: Baseline to 1 hour
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
Number analyzed (Participants) | 23 | 25 | 23
Participants | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of epidural placement until 1 hour after placement.
Description: In the 1% lidocaine group, 1 participant experienced an adverse event and was removed from analysis and 1 participant was removed because they did not receive the study drug. In the bupivacaine plus lidocaine group 2 patients were removed because they did not receive the study drug.
Arm/Group | 1% Lidocaine | 0.25% Bupivacaine | Bupivacaine Plus Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 0/25 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% Lidocaine (N=23) | 0.25% Bupivacaine (N=25) | Bupivacaine Plus Lidocaine (N=23)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT03103100/Prot_SAP_000.pdf